CLINICAL TRIAL: NCT05019417
Title: Glycerol-Phenylbutyrate Treatment in Children With MCT Mutation (Allan-Herndon- Dudley Syndrome)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Amnon Zung, Head of Pediatrics, Associate Clinical Profesor, the Hebrew University of Jerusalem, Israel, Kaplan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0089-19-KMC
Record Dates: First submitted 2021-07-01; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Monocarboxylate Transporter 8 Deficiency
Keywords: MCT8; Glycerol phenylbutyrate
MeSH Terms: conditions — Allan-Herndon-Dudley syndrome | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Glycerol phenylbutyrate treatment (Experimental): Name of the Investigational Medicinal product: Glycerol phenylbutyrate [GPB] (Ravicti oral liquid 1.1 gr/1 ml; manufacturer Horizon Pharma USA).
  Dosage of GPB will follow the dosage in use for children with urea cycle disorder.
  Initial dose: 5.0 gr (4.5 ml)/ meter square divided by three time a day. An escalating schedule dose of GPB will be used until normal serum T3 levels are reached.
  Initial dose: 5 gr/square meter body surface area (BSA). Second visit: 10 gr/square meter BSA
  The dose raising will be stopped if one of the following condition is reaches:
  1. Clinically significant side effects
  2. Reaching the PAA serum toxic threshold of 500 µg/ml
  3. Reaching the maximal dose of GPB that is in use in urea cycle disorder: 12.4 gr (11.2 ml)/ meter square BSA divided by three times a day.
  Duration of study: 4 months
  Interventions: Drug: Glycerol Phenylbutyrate 1100 MG/ML

INTERVENTIONS:
Drug: Glycerol Phenylbutyrate 1100 MG/ML — Daily adminisitraion of the study drug (three times a day) in escalting dose over 4 months
  Other Names: Ravicti (Horizon Pharma USA)

SUMMARY:
Rationale: Thyroid hormone (TH) is crucial for normal brain development. The transporter monocarboxlate transporter 8 (MCT8), located at various organs including brain neurons, is crucial for cellular transport of TH, mainly T3 . A defect in this transporter causes Allan-Herndon-Dudley syndrome (AHDS), which characterized by severe motor and cognitive retardation. Serum TH tests typically show low T4, high T3 and mildly elevated TSH. The neurological phenotype entails diminished TH transport into the brain. On the other hand, elevated serum T3 leads to hypermetabolic status in peripheral tissues. Subsequently, AHDS patients have a low body weight and muscle mass. Currently, no effective treatment is available. Over the last decade, several studies focused on the effect of T3 analogues, that their trans-membrane transport is not mediated by MCT8. Two analogues were studied: Diiodothyropropionic acid (DITPA) and tetraiodothyroacetic acid (Triac). Both agents have demonstrated improvement in serum TH levels (mainly T3 and TSH) but no change in the neurocognitive status of the patients.

Recently, several studies have demonstrated that sodium phenylbutyrate (PB) acting as a chaperon and increase the expression of MCT8 in the cell membrane. Subsequently, cells transfected with various mutations in MCT8 have shown remarkable improvement in T3 transport into the cytoplasm.

We hypothesize that treatment of AHDS patients with glycerol phenylbutyrate (GPB) will improve thyroid function and neurodevelopmental parameters and relieve symptoms resulting from toxic T3 levels in peripheral tissues.

Objective: To test safety and efficacy of PB treatment in AHDS patients.

Primary objectives:

To determine the effect of PB treatment on serum levels of TH.

Secondary objective:

1. To determine the effect of PB on T3-associated hyperthyroid state in peripheral tissues.
2. To determine the effects of PB treatment on the neurodevelopmental status. Study design: therapeutic prospective trial. Study population: Up to 6 AHDS patients with genetically proven ADHD. Intervention: all participants will receive an escalating dose of PB in the form of Glycerol-PB (commercial name Ravicti) until individual serum T3 levels have been normalized or dose limiting toxicities occur.

Duration of treatment: 12 months including the wash-out period of 1 month from the current Triac therapy

DETAILED DESCRIPTION:
1. Introduction and rationale

   Thyroid hormone (TH) is crucial for the development and metabolic state of virtually all tissues. TH signaling is regulated at the tissue level by intracellular conversion of the prohormone thyroxine (T4) to receptor-active 3,3',5-triiodothyronine (T3) or receptor-inactive 3,3',5'-triiodothyronine (rT3) by deiodinases. Since T3 receptors are located in the nucleus, TH transport across the plasma membrane is required for both TH metabolism and action. This process is facilitated by TH transporters, the most specific of which is monocarboxylate transporter 8 (MCT8) which is encoded by SLC16A2 gene located at chromosome X. MCT8 is critical for the transport of TH in a number of tissues, in particular the brain. Hemizygous mutations of MCT8 in males cause the Allan-Herndon-Dudley syndrome (AHDS), a severe neurodevelopmental disorder that is accompanied by abnormal TH levels.

   The neurological phenotype is characterized by severe neurodevelopmental retardation starting at the first few month of life. Initially, AHDS patients also have peripheral hypotonia but this usually progresses to spastic quadriplegia. Brain MRI of AHDS patients shows delayed myelination.

   The remarkable clinical spectrum of AHDS is probably derived from the defect in T3 entry in MCT8-expressing neurons and, thus, deprivation of TH in specific brain regions. The endocrine profile of patients with AHDS is characterized by moderately low T4, high T3 (usually more than twice the upper limit) and normal or mildly elevated TSH. The elevated serum T3 levels are toxic for peripheral tissues in which MCT8 is not important for TH transport, resulting in hyperthyroid symptoms such as low body weight, tachycardia, insomnia and muscle wasting. This peripheral phenotype is progressive with age.

   Currently, no effective therapy is available for AHDS patients. Over the last decade, the main research efforts focused on thyromimetic agents that are not relied on MCT8 but might enter the central nervous system (CNS) neurons through alternative membrane transporters. Studies in Mct8 KO mice with the T3 analog 3,5-diiodothyropropionic acid (DITPA) demonstrated T3-like effects in the brain and a decrease in serum T3 levels, which attenuated the thyrotoxic state of peripheral tissues. It should be emphasized however that although mice model mimics the thyroid function profile typical to AHDS, it has normal neurological development. This study prompted a study in 4 AHDS patients. DITPA treatment normalized the elevated serum levels of T3 and TSH, while T4 and rT3 levels were increased to normal lower range. There was improvement neither in neurodevelopmental functions nor in peripheral phenotype of the patients. Following the limited effects of DITPA treatment, an alternative thyromimetic agent was suggested: tetraiodothyroacetic acid (Triac [Tiratricol,Téatrois]). In a report of multicenter international studies published in The lancet Diabetes and Endocrinology (2019), escalating dose schedule of Triac yielded reduced levels of T3 to the normal range and similar reduction in T4 and TSH. Yet, there no improvement of motor and cognitive skills was observed.

   Over the last couple of years, a different potential therapeutic approach was suggested, by using chemical chaperons. The chaperons are molecules that are capable of altering stability of misfolded proteins and improving trafficking to the cell membrane. Several in-vitro studies have shown that the chemical chaperon sodium phenylbutyrate (PB) was able to rescue protein expression and the T3-transport function of various pathogenic MCT8 mutants. PB is routinely used in patients with urea-cycle disorder aiming at reducing their hyperammonemia, mainly in the form of glycerol-phenylbutyrate (GPB), a more palatable version of the drug.

   The investigators aim to perform a therapeutic study in order to evaluate the effect of GPB on the abnormal TH profile, the peripheral thyrotoxic effect of TH and the neurodevelopment status of AHDS patients with MCT8-confirmed mutations.
2. Objectives

The study will determine the effect of GPB on the abnormal TH profile, the peripheral thyrotoxic effect of TH and the neurodevelopment status of AHDS patients with MCT8-confirmed mutations.

Primary objective:

1) To evaluate the effect of GPB treatment on serum levels of T3 and other TH levels.

Secondary objective:

1. To determine the effect of GPB on hematological and biochemical parameters in AHDS patients and to recognize side effects of the treatment.
2. To determine the effect of GPB on T3-associated hyperthyroid state in peripheral tissues.
3. To determine the effects of GPB treatment on the neurodevelopmental status of the patients.

3. Study design

The investigators will perform a therapeutic prospective study in up to 6 AHDS with genetically-confirmed MCT8 mutation. Subjects will be recruited in our clinic and collaborating clinics. All participating patients will receive the investigational treatment glyceol-phenybuturate (GPB) in an individualized dose-escalation scheme for up to 4 months. There will be no control group or blinding.

Study population

1. Population AHDS patients with genetically-confirmed MCT8 mutations will be recruited in our clinic (The Pediatric Endocrinology Unit, Kaplan Medical Center, Rehovot, Israel) and collaborating clinics.
2. Inclusion criteria AHDS with characteristic clinical phenotype and with genetically confirmed mutation in the MCT8 gene SLC16A2.
3. Exclusion criteria

   * Inability to get the study medication GPB per-os (in cases without gastrotstomy)
   * Known contra-indication for GPB
   * Patients with AHDS but without confirmed mutation in the MCT8 gene

Treatment of subjects

1. Investigational product/treatment Name of the Investigational Medicinal product: Glycerol phenylbutirate [GPB] (Ravicti oral liquid 1.1 gr/1 ml; manufacturer Horizon Pharma USA).
2. Dosage of GPB will follow the dosage in use for children with urea cycle disorder.

   The initial dose will be 5.0 gr (4.5 ml)/ meter square divided by three time a day.

   An escalating schedule dose of GPB will be used until normal serum T3 levels are reached. The dose raising will be stopped if one of the following condition is reaches: 1. Clinically significant side effects 2. Reaching the PAA serum toxic threshold of 500 µg/ml 3. Reaching the maximal dose of GPB that is in use in urea cycle disorder: 12.4 gr (11.2 ml)/ meter square divided by three times a day. The maximal daily dose should not be above 19.0 gr (17.5 ml).

   Unlike urea cycle disorder where GPB dose is titrated by the serum ammonia levels, in AHDS patients ammonia levels are within normal limits, therefore, the titration should be based on the measurement of PAA in the serum, a derivative of GPB that is associated with neurotoxicity at high concentrations.
3. Safety profile of GPB Phenylbutirate is a pre-drug that undergoes hydrolysis by pancreatic lipases into phenylbutiric acid (PBA). Following first phase metabolism in the liver, PBA undergoes beta-oxidation into phenylacetic acid (PAA), the active metabolite of the drug. PAA then undergoes conjugation in the liver and the kidney into phenylacetylglutamin (PAGN) and secreted in the urine.

   Sodium phenylbutirate (NaPB) is currently in use for patients with hyperammonemia due to urea cycle disorders. Unlike sodium phenybutirate, the glycerol phenylbutirate (GPB) lacks taste and odor and is more palatable, therefore, it is preferred for therapeutic use. The potency ratio between the two derivatives is: NaPB x 0.86 = GPB. Based on the wide experience with GPB in children with urea cycle disorder, we will use this product in the study, with escalating dose that follow the therapeutic range in urea cycle disorder.

   The safety profile was evaluate in healthy adults and in patients with cirrhosis. The side effects of a single dose of GPB was evaluated in 24 healthy individuals and the effect of several doses in 8 healthy individuals and 24 patients with cirrhosis. By comparison to NaPB, the maximal concentrations of the metabolites of GPB were lower and appeared later. The degradation to PAGN was slower (as measured in urine). The degradation to PAGN in healthy individuals and patients with cirrhosis was similar. Side effects that were reported in this study were dizziness, headache and nausea. Hematological and biochemical parameters (including liver function tests) and coagulation factors were within normal limits. Similarly, no significant changes were recorded in the EKG. Since PAA is a GPB derived metabolite with neurotoxic effect, the toxic level of PAA was calculated and found to be much higher that the maximal serum concentration of PAA observed in this study.
4. Side effects

Common:

Skin : rash (10%) Reduced appetite (7%) GI tract: diarrhea (10%), vomiting (7%), abdominal pain, flatulence, dyspepsia Neurology: Dizziness (10%), headache (10%), weakness (7%)

Severe:

Neurotoxicity (dizziness, hypaucusis, dygeusia. These side effects were reported in association with high levels of PAA in the serum

Metabolic:

Reduced levels of branched-chain amino-acids: leucine, isoleucine, valine

Study protocol

1. A washout time of at least 4 weeks (without any medication such as Triac, DITPA or TH) will precede the initiation of the study.

   There are three clinic visits in the study, over 4 months:

   Initiation visit, 2 months, 4 months (final visit)
2. The following measurements and tests will be performed in every visit:

   Anthropometric measurements: height, weight, blood pressure, pulse, head circumference Neurological evaluation: A neurological examination will be deployed to assess the presence of hyperreflexia , primitive reflexes and hypertonia.

   Hyperreflexia will be assessed by the biceps, triceps, patellar and ankle tendon reflexes at both sides, and be scored on predefined scale Primitive reflexes: the following primitive reflexes will be evaluated: glabellar, snout, sucking, grasp and palmomental reflex.

   Hypertonia will be measured using the modified Ashworth scale in the upper (elbow) and lower (knee) extremities at both sides and be scored on a scale from 0 (no increase in muscle tone) to 4 (rigidity in both flexion and extension). Hypertonia will be defined as a score of >2 in at least one location at both sides of the body.

   Electrocardiogram for heart rate, PR length, QRS length, QT corrected value

   Blood tests:

   CBC (complete blood count) Chemistry: Na, K, ALT, AST, LDH, Alkaline phosphatase, GGT, urea, creatinine, total protein, albumin, uric acid, cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, calcium, phosphate, glucose, CPK Sex hormone binding globulin (SHBG) Ammonia Thyroid function tests: TSH, free T4 (FT4), total T4 (TT4), free T3 (FT3), thyroglobulin Serum amino acids profile Serum levels of phenylacetate (by mass spectrometry)
3. The following measurements will be performed only in the first and final visit:

   Gross motor function measure (GMFM) score sheet (GMFM-88) Bayley scales of infant development (BSID) III Adaptive behavior assessment system II (ABAS) for parents
4. Drug accountability: A record of study drug movement will be maintained for accountability purposes. In each visit, the legal guardian of the patients will be the empty cans of the study drug. The number of empty cans will be recorded.
5. Side effects: In each visit, a review of all adverse effect will be recorded. In addition, the legal guardians will receive a list of all adverse effects of the study drug, and will record adverse effects by day and hour between the clinic visits.

ELIGIBILITY:
Inclusion Criteria:

AHDS with characteristic clinical phenotype and with genetically confirmed mutation in the MCT8 gene SLC16A2.

Exclusion Criteria:

* Inability to get the study medication glycerol phenylbutyrate per-os (in cases without gastrotstomy)
* Known contra-indication for glycerol phenylbutyrate
* Patients without confirmed mutation in the MCT8 gene

Ages: 6 Months to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The disease is X-linked and basically appears only in males
Enrollment: 6 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Normalization of thyroid function test in response to glycerol phenylbutyrate | 4 months
  Serum free T4 (ng/dl), Serum total T4 (nmol/L), Serum free T3 (pg/ml), Serum TSH (microIU/ml), Serum thyroglobulin (ng.ml)

SECONDARY OUTCOMES:
The effect of glycerol phenybutyrat on hematological and biochemical parameters in patients | 4 months
  complete blood count, sex-hormone binding protein, chemistry, ammonia,
Height and weight gain in response to glycerol phenylbutyrate treatment | 4 months
  Body height (cm), Body weight (kg)
improvement in motor function in response to glycerol phenylbutyrate treatment | 4 months
  Gross motor function measure scoring outcome. Score range 0-264. Higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Zung, MD, Principal Investigator — Kaplan Medical Center, affiliated with the Hebrew University of Jerusalem, Israel
Locations (1):
- Pediatric Endocrinology Unit, Kapan Medical Center, Rehovot, Israel